CLINICAL TRIAL: NCT04631380
Title: A Double Blind, Controlled, Randomized, Prospective Study That Will Evaluate the Impact of Remote Intercession Prayer on the Clinical Evolution of Patients Diagnosed With COVID -19 in HCOR.
Brief Title: Prayer in Commbate to Corona Virus - Covid -19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRAYER-COVID19
Record Dates: First submitted 2020-08-04; First posted 2020-11-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Faith Healing

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE RANDOMIZED DOUBLE-BLIND STUDY
Who Masked: Participant
Masking Description: RAMDOMIZED DOBLE-BLINDING
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): THIS GROUP WILL RECEIVE THE PROTCOLL TREATMENT GIVEN TO PATIENTS COVID -POSITIVE TESTED.
- PRAYER (Experimental): THIS GROUP WILL RECEIVE THE SAME TREATMENT GIVEN TO THE CONTROL GROUP, PLUS PRAYERS BY THEOLOGIANS WHOSE PRAYERS INTERCEDE IN FAVOR OF THEIR PROMPT RECOVERY
  Interventions: Other: PRAYER

INTERVENTIONS:
Other: PRAYER — THE PRAYER GROUP WILL RECEIVE ABSOLUTELY THE SAME CARE AS THE CONTROL GROUP PLUS PRAYERS
  Other Names: INTERCESSORY PRAYER
  Arms: PRAYER

SUMMARY:
PATIENTS WHO ARE ADMITTED TO HOSPITALIZATION IN HCOR AND WHO HAVE THE CONFIRMED DIAGNOSIS OF CORONA VIRUS, WILL BE ASKED TO CONSENT TO PARTICIPATE IN THIS STUDY THAT INTENDS TO STUDY THE EFFECTIVENESS OF THE REMOTE INTERCESSION PRAYER IN COMBATING THIS DISEASE.

DETAILED DESCRIPTION:
PATIENTS WHO AGREE TO PARTICIPATE IN THE STUDY WILL BE SEPARATED INTO 2 GROUPS, THE INTERVENTION GROUP AND THE CONTROL GROUP.

THE IDENTITY OF THE PATIENTS WILL BE KEPT IN SECRET AND ONLY THEIR INITIALS WILL BE LISTED.

THE INTERVENTION GROUP WILL RECEIVE DAILY PRAYERS AND THE EVOLUTIONARY CLINICAL RESULTS OF THE TWO GROUPS WILL BE PURCHASED.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized in comun hospital rooms and intensive care units with confirmed COVID-19.

Exclusion Criteria:

* Patients admitted to the HCor emergency room, diagnosed with COVID-19 infection, however, without indication for hospitalization
* Patients admitted to the HCor emergency room, diagnosed with COVID-19 infection, however, without indication for hospitalization.
* Patients 18 years of age or older
* Patients with indication of palliative care and definition of terminality at hospital admission
* Patients who voluntarily choose not to participate in the study at the time of the • presentation of the Informed Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
DEATH OR RECOVERY | 60 DAYS
  WE WILL EVALUATE DEATHS OR HOSPITAL DISCHARGE

SECONDARY OUTCOMES:
NEED FOR MECHANICAL VENTILATION | 60 DAYS
  NEED FOR MECHANICAL VENTILATION
TIME OF REMAINED INTUBATED | 60 DAYS
  TIME OF REMAINED INTUBATED
LENGTH OF STAY IN ICU | 60 DAYS
  LENGTH OF STAY IN ICU
TIME OF STAY HOSPITALIZED | 60 DAYS
  TIME OF STAY HOSPITALIZED
Occurrence of clinical complications. | 60 DAYS
  Occurrence of clinical complications that were not included before diagnostic confirmation and that may be related to covid infection.

CONTACTS AND LOCATIONS:
Overall Officials: NATHAN V SOUBIHE JR, Principal Investigator — Hospital do Coracao
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
They will not

REFERENCES:
- [Background] Hettiaratchy S, Hemsley C. Effect of retroactive intercessory prayer. Paper proves power of statistics, not prayer. BMJ. 2002 Apr 27;324(7344):1037; author reply 1038-9. No abstract available. PMID 11977259
- [Background] Harris WS, Gowda M, Kolb JW, Strychacz CP, Vacek JL, Jones PG, Forker A, O'Keefe JH, McCallister BD. A randomized, controlled trial of the effects of remote, intercessory prayer on outcomes in patients admitted to the coronary care unit. Arch Intern Med. 1999 Oct 25;159(19):2273-8. doi: 10.1001/archinte.159.19.2273. PMID 10547166
- [Background] Hoover DR, Margolick JB. Questions on the design and findings of a randomized, controlled trial of the effects of remote, intercessory prayer on outcomes in patients admitted to the coronary care unit. Arch Intern Med. 2000 Jun 26;160(12):1875-6; author reply 1877-8. doi: 10.1001/archinte.160.12.1875-b. No abstract available. PMID 10871995
- [Background] Radin D, Schlitz M, Baur C. Distant Healing Intention Therapies: An Overview of the Scientific Evidence. Glob Adv Health Med. 2015 Nov;4(Suppl):67-71. doi: 10.7453/gahmj.2015.012.suppl. Epub 2015 Nov 1. PMID 26665044
- [Background] Bleich A. [Intercessory prayer for health: a matter of faith, science or both]. Harefuah. 2002 Jun;141(6):522-3. No abstract available. Hebrew. PMID 12119766